CLINICAL TRIAL: NCT06979024
Title: A Registered Observational Cohort Study of Myotonic Dystrophy Type 1
Status: Enrolling by invitation | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA,ECFAH of FMU [2015]084-2; 8240063043 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2025-04-28; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
Keywords: Myotonic Dystrophy Type 1; Tandem repeat
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples stored in -80
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of Patients with Myotonic Dystrophy Type 1 (DM1): This cohort includes patients with Myotonic Dystrophy Type 1 (DM1), focusing on clinical observations to understand the natural progression of the disease. Observations cover changes in muscle function, respiratory capacity, cardiac health, and quality of life. Additionally, third-generation sequencing is used to determine repeat numbers, exploring the relationship between repeat expansion and clinical phenotypes. These insights aim to identify biomarkers of disease progression and provide foundational data for future therapeutic research.
  Interventions: Genetic: Triplet-primed PCR or Long-read sequencing

INTERVENTIONS:
Genetic: Triplet-primed PCR or Long-read sequencing — This study involves long-read sequencing in patients with Myotonic Dystrophy Type 1 (DM1) to identify specific motifs, determine the range of repeat numbers, and assess the presence of interruptions in the CTG repeat sequence. The aim is to gain insights into the genetic variability and its clinical implications in DM1.

SUMMARY:
Myotonic dystrophy type 1 (DM1) is the most common form of muscular dystrophy.There is little phenotype and genetic data for Chinese DM1 patients. The data to be collected is intended to fill this gap and provide complementary data

DETAILED DESCRIPTION:
Myotonic dystrophy 1 (DM1) is an autosomal, dominantly inherited neuromuscular disorder characterized by skeletal muscle weakness, myotonia, cardiac conduction abnormalities, cataracts, and other abnormalities. The China DM1 patient registry is a nationwide, population-based, non-interventional, observational cohort clinical study of all age groups of genetically-confirmed DM1 patients from families (with at least 1 affected member), collecting data retrospectively at study entry and prospectively during follow up. Currently, there is limited phenotype and genotype data available for DM1 patients with Chinese Han ethnicity. Therefore, the data to be collected is intended to fill this gap and provide complementary data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of all ages at baseline
* Subjects, with or without symptoms, with DM1 genetic confirmation through triplet-primed PCR or long-read sequencing
* Unrelated healthy controls

Exclusion Criteria:

* Decline to participate
* Other neuromuscular disease (such as Limb-girdle muscular dystrophy or Oculopharyngodistal Myopathy)
* Serious systemic illness (such as heart, liver, kidney disease or major mental illness)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All genetically-confirmed DM1 patients from families (with at least 1 affected member) in China, irrespective of age. The CTG repeats presented at least 50 repeats in DMPK gene, the diagnosis of which was performed at Fujian Neuromedical Center (FNMC), the clinical genetic test hospital for DM1 in China to employ triplet-primed PCR or long-read sequencing technology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Triplet-primed PCR or Long-read sequencing | Baseline
  Genetic test of triplet-primed PCR or long-read sequencing is performed for these clinical suspected DM1 patients on the basis of the family as a whole. Eligible participants are genetically confirmed patients With CTG repeats >50 in DMPK gene.
Muscle Impairment Rating Scale (MIRS) | Baseline through study completion (an average of 1 year)
  This scale evaluates muscular impairment severity according to an ordinal 5-point scale as follows: (1) no muscular impairment, (2) minimal signs, (3) distal weakness, (4) mild to moderate proximal weakness, and (5) severe proximal weakness.
The modified Medical Research Council (MRC) scale | Baseline through study completion (an average of 1 year)
  The modified Medical Research Council (MRC) scale is used to assess numerically the muscle strength of DM1 participants. Firstly, muscles are tested bilaterally (when applicable) in standardized positions with manual muscle testing (MMT) scores. Then, MMT scores are converted to calculable data of the modified MRC scale.

SECONDARY OUTCOMES:
Changes in 6-Minute Walk Test | Baseline through study completion (an average of 1 year)
  The 6-Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered in 6 minutes serves as the outcome for comparing changes in performance capacity.
Changes in 10 Metre Walk Test (10MWT) | Baseline through study completion (an average of 1 year)
  The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
Requests for IPD will be evaluated on a case-by-case basis.